CLINICAL TRIAL: NCT04048551
Title: The PrEPARE Project: Prevention, Empowering, and Protecting Young Women in South Africa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RTI International (Other)
Collaborators: Setshaba Research Centre (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: R01HD094629 (NIH)
Record Dates: First submitted 2019-05-28; First posted 2019-08-07 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: HIV Prevention
Keywords: PrEP (Pre-exposure Prophylaxis); HIV (Human Immunodeficiency Virus); Adolescent Girls and Young Women (AGYW); Stigma and Discrimination (S&D); Gender-based violence (GBV); Substance use
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Social Stigma; Substance-Related Disorders | interventions — N-(4'-fluorobutyrophenone)-4-(4-chlorophenyl)pyridinium

STUDY DESIGN:
Intervention Model Description: This is a cluster randomized trial that utilizes a 2 x 2 factorial design to assess the impact of S&D reduction training and the YWHC intervention, resulting in four study conditions: (1) Clinic S&D reduction training + PrEP/SRH + YWHC, (2) Clinic S&D reduction training + PrEP/SRH only, (3) No Clinic S&D reduction training +PrEP/SRH + YWHC, (4) No Clinic S&D reduction training + PrEP/SRH only. The researchers will examine two primary endpoints: (1) the proportion of AGYW who are ready to uptake and initiate PrEP and SRH services; and, (2) the differences in levels of PrEP adherence between each intervention condition and the standard of care comparison at 3-, 6- and 9-month follow-up.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- No S&D Reduction Training; PrEP and SRH only (No Intervention): Arm 1 does not receive stigma and discrimination (S&D) reduction training to clinic staff, but provides PrEP (pre-exposure prophylaxis) and SRH (sexual and reproductive health) services to AGYW (adolescent girls and young women).
- No S&D Reduction Training; PrEP and SRH + YWHC (Experimental): Arm 2 does not receive stigma and discrimination (S&D) reduction training to clinic staff, but provides PrEP (pre-exposure prophylaxis), SRH (sexual and reproductive health) services, and YWHC (Young Women's Health CoOp) to AGYW (adolescent girls and young women).
  Interventions: Behavioral: Young Women's Health CoOp (YWHC)
- S&D Reduction Training; PrEP and SRH only (Active Comparator): Arm 3 receives stigma and discrimination (S&D) reduction training to clinic staff and provides PrEP (pre-exposure prophylaxis) and SRH (sexual and reproductive health) services to AGYW (adolescent girls and young women).
  Interventions: Behavioral: Modified Health Policy Project (HPP) HIV-Stigma and Discrimination Reduction Training Curriculum
- S&D Reduction Training; PrEP, SRH + YWHC (Experimental): Arm 4 receives stigma and discrimination (S&D) reduction training to clinic staff and provides PrEP (pre-exposure prophylaxis), SRH (sexual and reproductive health) services, and YWHC (Young Women's Health CoOp) to AGYW (adolescent girls and young women).
  Interventions: Behavioral: Modified Health Policy Project (HPP) HIV-Stigma and Discrimination Reduction Training Curriculum; Behavioral: Young Women's Health CoOp (YWHC)

INTERVENTIONS:
Behavioral: Modified Health Policy Project (HPP) HIV-Stigma and Discrimination Reduction Training Curriculum — The Health Policy Project (HPP) training curriculum provides participatory training modules that address three key actionable drivers of HIV-stigma. The HPP curriculum was adapted through participatory workshops with key stakeholders representing clinics, study staff, and adolescent girls and young women (AGYW) and other formative activities. The training is a whole-site training to address barriers to accessing clinical services by AGYW. Consequently, staff at all levels (clinical and nonclinical) will be trained on stigma and discrimination as it relates to AGYW in order to reduce stigma-related barriers to healthcare and increase uptake of PrEP and sexual and reproductive health services among AGYW.
  Arms: S&D Reduction Training; PrEP and SRH only; S&D Reduction Training; PrEP, SRH + YWHC
Behavioral: Young Women's Health CoOp (YWHC) — In this study, researchers adapted the Young Women's Health CoOp (YWHC) evidence-based empowerment intervention that addresses issues of gender-based violence (GBV), substance use, and sexual risk to include information about PrEP (pre-exposure prophylaxis) and sexual and reproductive health. AGYW will be provided with comprehensive information and will engage in activities that seek to reduce HIV risk factors and increase PrEP readiness, uptake and adherence.
  Arms: No S&D Reduction Training; PrEP and SRH + YWHC; S&D Reduction Training; PrEP, SRH + YWHC

SUMMARY:
The project seeks to determine whether implementing a multilevel, woman-focused intervention, the Young Women's Health CoOp (YWHC), for pre-exposure prophylaxis (PrEP) readiness, uptake, and adherence is a viable complement to the HIV prevention plan for the Government of South Africa. Specifically, this project aims to: increase uptake, of sexual and reproductive health (SRH) services and readiness and uptake of PrEP among adolescent girls and young women (AGYW) aged 16 to 24 who engage in high-risk sexual behaviors; and reduce their barriers to accessing SRH services by addressing and reducing stigma and discrimination (S&D) in clinics.

DETAILED DESCRIPTION:
The researchers propose a cluster randomized trial with a factorial design to evaluate the efficacy of a multi-level intervention that addresses stigma in accessing healthcare, social support, and individual risk behaviors of adolescent girls and young women (AGYW) in South Africa. The researchers engaged stakeholders from the Department of Health, a Community Collaborative Board (CCB), and a Youth Advisory Board (YAB) to inform the adaptation of the evidence-based empowerment intervention, the Women's Health CoOp (WHC)-which addresses gender-based violence (GBV), substance use, and sexual risk-to address sexual and reproductive health (SRH) and pre-exposure prophylaxis (PrEP) readiness, uptake and adherence. Through engagement with stakeholders, the researchers also adapted a stigma and discrimination (S&D) reduction training curriculum for clinic staff.

The project plans to increase uptake of SRH services, and PrEP readiness, uptake and adherence among AGYW aged 16 to 24 who engage in high-risk sex. The investigators plan to conduct this through a multilevel HIV prevention strategy that addresses S&D in AGYW accessing healthcare, social support, and individual risk behaviors. This cluster randomized trial with a factorial design will be conducted across 12 clinics in Pretoria.

The aims of this study are (1) To engage stakeholders, the Community Collaborative Board (CCB), and the Youth Advisory Board (YAB) in adapting the Women's Health CoOp (WHC) and stigma and discrimination (S&D) reduction training, in the Pretoria area during a formative stage.

(2) To evaluate the impact of training on S&D among healthcare staff on the use of HIV and reproductive health services by adolescent girls and young women (AGYW), including pre-exposure prophylaxis (PrEP), and staff attitudes and behaviors toward AGYW at 4- and 8-month follow-up.

(3) To test the efficacy of a multilevel strategy that addresses structural (stigma and discrimination), interpersonal (social support), and individual (personal agency, substance use, and gender-based violence [GBV]) factors on PrEP readiness and uptake, and adherence (primary outcomes) and condom use, GBV, substance use, and HIV incidence (secondary) at 3-, 6-, and 9-month follow-up among vulnerable AGYW.

ELIGIBILITY:
Inclusion Criteria:

* HIV negative
* identify as female;
* aged 16-24;
* have had condomless sex in the past 3 months with a male partner;
* not be currently pregnant and not want to get pregnant for the next year;
* interested in taking PrEP;
* not having previously participated in the formative phase of the study;
* have not previously and not currently participating in any other PrEP-related demonstration project or research study;
* not previously or not currently participating in any other HIV study in Tshwane;
* lives in one of the target communities;
* not on multidrug-resistant tuberculosis (MDR-TB) treatment;
* intends to stay in the Tshwane district for the next 12 months;
* agrees to provide contact information;
* be willing to undergo rapid HIV testing;
* be willing to undergo pregnancy testing.

Exclusion Criteria:

-

Ages: 16 Years to 24 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 802 (Actual)
Dates: Start 2019-04-04 (Actual); Primary Completion 2022-06-23 (Actual); Study Completion 2022-06-23 (Actual)

PRIMARY OUTCOMES:
Health Clinic-Level Outcome: Level of Health Clinic Stigma and Discrimination | Baseline
  Staff surveys that are modified from the Health Policy Project survey will be used to measure healthcare staffs' attitudes toward sexually active AGYW; the overall clinic environment; observed discrimination and stigmatizing behaviors toward AGYW. Greater values indicate higher levels of health clinic stigma and discrimination.
Health Clinic-Level Outcome: Level of Health Clinic Stigma and Discrimination | 4 months
  Staff surveys that are modified from the Health Policy Project survey will be used to measure healthcare staffs' attitudes toward sexually active AGYW; the overall clinic environment; observed discrimination and stigmatizing behaviors toward AGYW. Greater values indicate higher levels of health clinic stigma and discrimination.
Health Clinic-Level Outcome: Level of Health Clinic Stigma and Discrimination | 8 months
  Staff surveys that are modified from the Health Policy Project survey will be used to measure healthcare staffs' attitudes toward sexually active AGYW; the overall clinic environment; observed discrimination and stigmatizing behaviors toward AGYW. Greater values indicate higher levels of health clinic stigma and discrimination.
Health Clinic-Level Outcome: The Number of AGYW who Uptake HIV and SRH services, including PrEP | Baseline
  A clinic audit, including a review of administrative data, will be conducted to assess the number of AGYW who uptake HIV and sexual and reproductive health services, including PrEP in each clinic.
Health Clinic-Level Outcome: The Number of AGYW who Uptake HIV and SRH services, including PrEP | 4 months
  A clinic audit, including a review of administrative data, will be conducted to assess the number of AGYW who uptake HIV and sexual and reproductive health services, including PrEP in each clinic.
Health Clinic-Level Outcome: The Number of AGYW who Uptake HIV and SRH services, including PrEP | 8 months
  A clinic audit, including a review of administrative data, will be conducted to assess the number of AGYW who uptake HIV and sexual and reproductive health services, including PrEP in each clinic.
AGYW Participant Self-Report: The Level of PrEP Readiness among AGYW | Baseline
  Self-report responses to a modified scale from the HIV Prevention Trials Network (HPTN) 082 trial and single item measures developed for this study and from the adapted Risk Behavior Assessment (RBA) questionnaires will be used to assess the extent to which AGYW are ready to initiate PrEP. Greater values indicate higher levels of PrEP readiness.
AGYW Participant Self-Report: The Level of PrEP Readiness among AGYW | 3 months
  Self-report responses to a modified scale from the HIV Prevention Trials Network (HPTN) 082 trial and single item measures from the adapted Risk Behavior Assessment (RBA) questionnaires will be used to assess the extent to which AGYW are ready to initiate PrEP. Greater values indicate higher levels of PrEP readiness.
AGYW Participant Self-Report: The Level of PrEP Readiness among AGYW | 6 months
  Self-report responses to a modified scale from the HIV Prevention Trials Network (HPTN) 082 trial and single item measures from the adapted Risk Behavior Assessment (RBA) questionnaires will be used to assess the extent to which AGYW are ready to initiate PrEP. Greater values indicate higher levels of PrEP readiness.
AGYW Participant Self-Report: The Level of PrEP Readiness among AGYW | 9 months
  Self-report responses to a modified scale from the HIV Prevention Trials Network (HPTN) 082 trial and single item measures from the adapted Risk Behavior Assessment (RBA) questionnaires will be used to assess the extent to which AGYW are ready to initiate PrEP. Greater values indicate higher levels of PrEP readiness.
AGYW Participant Self-Report: PrEP Uptake and Adherence among AGYW | 3 months
  Self-report responses to a modified scale from Microbicide Trials Network Studies (MTN) and single item measures from the adapted Risk Behavior Assessment (RBA) questionnaires will be used to assess if AGYW initiated PrEP. Self-report responses on the AGYW questionnaire adapted from previous research will be used to assess PrEP adherence, including past 30-day use, and patterns of use, persistence and discontinuation.
AGYW Participant Self-Report: PrEP Uptake and Adherence among AGYW | 6 months
  Self-report responses to a modified scale from Microbicide Trials Network Studies (MTN) and single item measures from the adapted Risk Behavior Assessment (RBA) questionnaires will be used to assess if AGYW initiated PrEP. Self-report responses on the AGYW questionnaire adapted from previous research will be used to assess PrEP adherence, including past 30-day use, and patterns of use, persistence and discontinuation.
AGYW Participant Self-Report: PrEP Uptake and Adherence among AGYW | 9 months
  Self-report responses to a modified scale from Microbicide Trials Network Studies (MTN) and single item measures from the adapted Risk Behavior Assessment (RBA) questionnaires will be used to assess if AGYW initiated PrEP. Self-report responses on the AGYW questionnaire adapted from previous research will be used to assess PrEP adherence, including past 30-day use, and patterns of use, persistence and discontinuation.
AGYW Biological Outcome: Adherence to PrEP | 3 months
  Dried blood spot samples will be used to measure the amount of drug (Tenofovir-diphosphate) concentration in AGYW's blood to assess PrEP adherence.
AGYW Biological Outcome: Adherence to PrEP | 6 months
  Dried blood spot samples will be used to measure the amount of drug (Tenofovir-diphosphate) concentration in AGYW's blood to assess PrEP adherence.
AGYW Biological Outcome: Adherence to PrEP | 9 months
  Dried blood spot samples will be used to measure the amount of drug (Tenofovir-diphosphate) concentration in AGYW's blood to assess PrEP adherence.
AGYW Participant Self-Report: Sexual and Reproductive Health Uptake among AGYW | 3 months
  Self-report responses on the single item measures from the adapted Risk Behavior Assessment (RBA) questionnaires will be used to assess if AGYW initiated SRH services.
AGYW Participant Self-Report: Sexual and Reproductive Health Uptake among AGYW | 6 months
  Self-report responses on the single item measures from the adapted Risk Behavior Assessment (RBA) questionnaires will be used to assess if AGYW initiated SRH services.
AGYW Participant Self-Report: Sexual and Reproductive Health Uptake among AGYW | 9 months
  Self-report responses on the single item measures from the adapted Risk Behavior Assessment (RBA) questionnaires will be used to assess if AGYW initiated SRH services.

SECONDARY OUTCOMES:
AGYW Participant Self-Report: Frequency of Drug Use | Baseline
  Self-report responses on the AGYW questionnaire adapted from previous research will be used to assess the frequency of drug (e.g, methamphetamine) use and injecting.
AGYW Participant Self-Report: Frequency of Drug Use | 3 months
  Self-report responses on the AGYW questionnaire adapted from previous research will be used to assess the frequency of drug (e.g, methamphetamine) use and injecting.
AGYW Participant Self-Report: Frequency of Drug Use | 6 months
  Self-report responses on the AGYW questionnaire adapted from previous research will be used to assess the frequency of drug (e.g, methamphetamine) use and injecting..
AGYW Participant Self-Report: Frequency of Drug Use | 9 months
  Self-report responses on the AGYW questionnaire adapted from previous research will be used to assess the frequency of drug (e.g, methamphetamine) use and injecting.
AGYW Participant Self-Report: Frequency of Alcohol Use | Baseline
  Self-report responses on the AGYW questionnaire adapted from previous research will be used to assess the number of days of alcohol consumption and the number of days of problematic (4+) alcohol consumption.
AGYW Participant Self-Report: Frequency of Alcohol Use | 3 months
  Self-report responses on the AGYW questionnaire adapted from previous research will be used to assess the number of days of alcohol consumption and the number of days of problematic (4+) alcohol consumption
AGYW Participant Self-Report: Frequency of Alcohol Use | 6 months
  Self-report responses on the AGYW questionnaire adapted from previous research will be used to assess the number of days of alcohol consumption and the number of days of problematic (4+) alcohol consumption
AGYW Participant Self-Report: Frequency of Alcohol Use | 9 months
  Self-report responses on the AGYW questionnaire adapted from previous research will be used to assess the number of days of alcohol consumption and the number of days of problematic (4+) alcohol consumption.
AGYW Participant Self-Report: Frequency of Combining Drugs and Alcohol Use | baseline
  Self-report responses on the AGYW questionnaire adapted from previous research will be used to assess the frequency of combining drugs with alcohol.
AGYW Participant Self-Report: Frequency of Combining Drugs and Alcohol Use | 3 months
  Self-report responses on the AGYW questionnaire adapted from previous research will be used to assess the frequency of combining drugs with alcohol.
AGYW Participant Self-Report: Frequency of Combining Drugs and Alcohol Use | 6 Months
  Self-report responses on the AGYW questionnaire adapted from previous research will be used to assess the frequency of combining drugs with alcohol.
AGYW Participant Self-Report: Frequency of Combining Drugs and Alcohol Use | 9 months
  Self-report responses on the AGYW questionnaire adapted from previous research will be used to assess the frequency of combining drugs with alcohol.
AGYW Participant Self-Report: Frequency of Condom Use | Baseline
  Self-report responses on single-item questions will be used to assess condom use. Condom use will be calculated as a count and percentage (based on the total number of acts and the numbers of acts with a condom). Lower percentage values indicate less frequent condom use. For the count variable, greater values indicate more acts of sex without a condom.
AGYW Participant Self-Report: Frequency of Condom Use | 3 months
  Self-report responses on single-item questions will be used to assess condom use. Condom use will be calculated as a count and percentage (based on the total number of acts and the numbers of acts with a condom). Lower percentage values indicate less frequent condom use. For the count variable, greater values indicate more acts of sex without a condom.
AGYW Participant Self-Report: Frequency of Condom Use | 6 months
  Self-report responses on single-item questions will be used to assess condom use. Condom use will be calculated as a count and percentage (based on the total number of acts and the numbers of acts with a condom). Lower percentage values indicate less frequent condom use. For the count variable, greater values indicate more acts of sex without a condom.
AGYW Participant Self-Report: Frequency of Condom Use | 9 months
  Self-report responses on single-item questions will be used to assess condom use. Condom use will be calculated as a count and percentage (based on the total number of acts and the numbers of acts with a condom). Lower percentage values indicate less frequent condom use. For the count variable, greater values indicate more acts of sex without a condom.
AGYW Participant Self-Report: Frequency of Alcohol and Other Drug Use Prior to or During Sex | Baseline
  Self-report responses on single-item questions from the Pretoria Risk Behavior Assessment will be used to assess engagement in alcohol and other drug use prior to or during sex.
AGYW Participant Self-Report: Frequency of Alcohol and Other Drug Use Prior to or During Sex | 3 months
  Self-report responses on single-item questions from the Pretoria Risk Behavior Assessment will be used to assess engagement in alcohol and other drug use prior to or during sex.
AGYW Participant Self-Report: Frequency of Alcohol and Other Drug Use Prior to or During Sex | 6 months
  Self-report responses on single-item questions from the Pretoria Risk Behavior Assessment will be used to assess engagement in alcohol and other drug use prior to or during sex.
AGYW Participant Self-Report: Frequency of Alcohol and Other Drug Use Prior to or During Sex | 9 months
  Self-report responses on single-item questions from the Pretoria Risk Behavior Assessment will be used to assess engagement in alcohol and other drug use prior to or during sex.
AGYW Participant Self-Report: Number of Other Sex Partners | Baseline
  Self-report responses on the AGYW questionnaire adapted from previous research will be used to assess the number of other sex partners among AGYW.
AGYW Participant Self-Report: Number of Other Sex Partners | 3 months
  Self-report responses on the AGYW questionnaire adapted from previous research will be used to assess the number of other sex partners among AGYW.
AGYW Participant Self-Report: Number of Other Sex Partners | 6 months
  Self-report responses on the AGYW questionnaire adapted from previous research will be used to assess the number of other sex partners among AGYW.
AGYW Participant Self-Report: Number of Other Sex Partners | 9 months
  Self-report responses on the AGYW questionnaire adapted from previous research will be used to assess the number of other sex partners among AGYW.
AGYW Participant Self-Report: Engagement in Sex Trading | Baseline
  Self-report responses on single-item measures modified from the Pretoria Risk Behavior Assessment (PRBA) will be used to assess whether participants engaged in trading sex for money or other things.
AGYW Participant Self-Report: Engagement in Sex Trading | 3 months
  Self-report responses on single-item measures modified from the Pretoria Risk Behavior Assessment (PRBA) will be used to assess whether participants engaged in trading sex for money or other things.
AGYW Participant Self-Report: Engagement in Sex Trading | 6 months
  Self-report responses on single-item measures modified from the Pretoria Risk Behavior Assessment (PRBA) will be used to assess whether participants engaged in trading sex for money or other things.
AGYW Participant Self-Report: Engagement in Sex Trading | 9 months
  Self-report responses on single-item measures modified from the Pretoria Risk Behavior Assessment (PRBA) will be used to assess whether participants engaged in trading sex for money or other things.
AGYW Participant Self- Report: Engagement with multiple sex partners (≥ 2 partners) | Baseline
  Self-report responses on the AGYW questionnaire adapted from previous research will be used to assess engagement with more than one sex partner in the past 3 months.
AGYW Participant Self- Report: Engagement with multiple sex partners (≥ 2 partners) | 3 months
  Self-report responses on the AGYW questionnaire adapted from previous research will be used to assess engagement with more than one sex partner in the past 3 months.
AGYW Participant Self- Report: Engagement with multiple sex partners (≥ 2 partners) | 6months
  Self-report responses on the AGYW questionnaire adapted from previous research will be used to assess engagement with more than one sex partner in the past 3 months.
AGYW Participant Self- Report: Engagement with multiple sex partners (≥ 2 partners) | 9 months
  Self-report responses on the AGYW questionnaire adapted from previous research will be used to assess engagement with more than one sex partner in the past 3 months.
AGYW Participant Self-Report: Use of Contraception | Baseline
  Self-report responses on single-item measures will be used to assess use of contraception and types of contraception among AGYW.
AGYW Participant Self-Report: Use of Contraception | 3 months
  Self-report responses on single-item measures will be used to assess use of contraception and types of contraception among AGYW.
AGYW Participant Self-Report: Use of Contraception | 6 months
  Self-report responses on single-item measures will be used to assess use of contraception and types of contraception among AGYW.
AGYW Participant Self-Report: Use of Contraception | 9 months
  Self-report responses on single-item measures will be used to assess use of contraception and types of contraception among AGYW.
Medical Record: Use of Contraception | Through study completion, an average of nine months
  Clinical medical record will be used to assess contraception and contraception type among AGYW.
AGYW Participant Self-Report: Level of Perception of HIV Risk | Baseline
  Self-report responses on single-item questions will be used to assess the extent to which AGYW perceive themselves as at risk for HIV infection. Higher levels indicate greater perceived HIV risk.
AGYW Participant Self-Report: Level of Perception of HIV Risk | 3 months
  Self-report responses on single-item questions will be used to assess the extent to which AGYW perceive themselves as at risk for HIV infection. Higher levels indicate greater perceived HIV risk.
AGYW Participant Self-Report: Level of Perception of HIV Risk | 6 months
  Self-report responses on single-item questions will be used to assess the extent to which AGYW perceive themselves as at risk for HIV infection. Higher levels indicate greater perceived HIV risk.
AGYW Participant Self- Report; Level of Perception of HIV Risk | 9 months
  Self-report responses on single-item questions will be used to assess the extent to which AGYW perceive themselves as at risk for HIV infection. Higher levels indicate greater perceived HIV risk.
AGYW Participant Self-Report: The Frequency of Experienced Stigma | Baseline
  Self-report responses on the AGYW questionnaire adapted from previous research will be used to assess the frequency of experiencing stigma or discrimination from clinic staff or community members among AGYW.
  .
AGYW Participant Self-Report: The Frequency of Experienced Stigma | 3 months
  Self-report responses on the AGYW questionnaire adapted from previous research will be used to assess the frequency of experiencing stigma or discrimination from clinic staff or community members among AGYW.
  .
AGYW Participant Self-Report: The Frequency of Experienced Stigma | 6 months
  Self-report responses on the AGYW questionnaire adapted from previous research will be used to assess the frequency of experiencing stigma or discrimination from clinic staff or community members among AGYW.
AGYW Participant Self-Report: The Frequency of Experienced Stigma | 9 months
  Self-report responses on the AGYW questionnaire adapted from previous research will be used to assess the frequency of experiencing stigma or discrimination from clinic staff or community members among AGYW.
AGYW Participant Self-Report: The Level of Anticipated Stigma | Baseline
  Self-report responses on single-item questions and multiple-item scales developed from the formative research study activities will be used to assess the extent to which AGYW anticipate stigma or discrimination from clinic staff or community members. Higher values indicate greater levels of anticipated stigma.
AGYW Participant Self-Report: The Level of Anticipated Stigma | 3 months
  Self-report responses on single-item questions and multiple-item scales developed from the formative research study activities will be used to assess the extent to which AGYW anticipate stigma or discrimination from clinic staff or community members. Higher values indicate greater levels of anticipated stigma.
AGYW Participant Self-Report: The Level of Anticipated Stigma | 6 months
  Self-report responses on single-item questions and multiple-item scales developed from the formative research study activities will be used to assess the extent to which AGYW anticipate stigma or discrimination from clinic staff or community members. Higher values indicate greater levels of anticipated stigma.
AGYW Participant Self-Report: The Level of Anticipated Stigma | 9 months
  Self-report responses on single-item questions and multiple-item scales developed from the formative research study activities will be used to assess the extent to which AGYW anticipate stigma or discrimination from clinic staff or community members. Higher values indicate greater levels of anticipated stigma.
  .
AGYW Participant Self-Report: The Frequency of Observed Stigma | Baseline
  Self-report responses on the AGYW questionnaire adapted from previous research will be used to the assess the frequency that AGYW have witnessed stigma or discrimination from clinic staff or community members toward sexually active AGYW.
AGYW Participant Self-Report: The Frequency of Observed Stigma | 3 months
  Self-report responses on the AGYW questionnaire adapted from previous research will be used to the assess the frequency that AGYW have witnessed stigma or discrimination from clinic staff or community members toward sexually active AGYW.
AGYW Participant Self-Report: The Frequency of Observed Stigma | 6 months
  Self-report responses on the AGYW questionnaire adapted from previous research will be used to the assess the frequency that AGYW have witnessed stigma or discrimination from clinic staff or community members toward sexually active AGYW.
AGYW Participant Self-Report: The Frequency of Observed Stigma | 9 months
  Self-report responses on the AGYW questionnaire adapted from previous research will be used to the assess the frequency that AGYW have witnessed stigma or discrimination from clinic staff or community members toward sexually active AGYW.

CONTACTS AND LOCATIONS:
Overall Officials: Felicia Browne, ScD, Principal Investigator — RTI International
Locations (1):
- Setshaba Research Centre, Soshanguve, South Africa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wechsberg WM, Browne FA, Ndirangu J, Bonner CP, Minnis AM, Nyblade L, Speizer IS, Howard BN, Myers B, Ahmed K. The PrEPARE Pretoria Project: protocol for a cluster-randomized factorial-design trial to prevent HIV with PrEP among adolescent girls and young women in Tshwane, South Africa. BMC Public Health. 2020 Sep 15;20(1):1403. doi: 10.1186/s12889-020-09458-y. PMID 32933510